CLINICAL TRIAL: NCT02303379
Title: Effects of Different Endurance Training Protocols on Physical Performance in Cardiac Patients
Brief Title: Different Endurance Training Protocols in Cardiac Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paracelsus Medical University (Other)
Responsible Party: Principal Investigator, Prof. Josef Niebauer M.D., Ph.D., MBA, Head of institute, Paracelsus Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UISM-8
Record Dates: First submitted 2014-11-25; First posted 2014-11-27 (Estimated); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Coronary Artery Disease
Keywords: Training Protocol; Cardiac Rehabilitation; High-Intensity Interval Training; Continuous Training; Pyramid Training; Physical Performance
MeSH Terms: conditions — Coronary Artery Disease | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Continuous Endurance training (Active Comparator): Endurance training with constant work load 31min at 65-75% maximal heart rate (HRmax)
  Interventions: Other: Pyramid Training; Other: High-intensity interval training
- Pyramid Training (Experimental): One pyramid consists of 8 one-minute blocks. Those are grouped starting with one block of 70-75% HRmax, followed by one block at 75-80% HRmax and another one at 80-85% HRmax. The top of the pyramid are 2 blocks of 85-90% HRmax. Intensity is lowered afterwards with one block of 80-85% HRmax, followed by one block at 75-80% HRmax and last one at 70-75% HRmax. Two more pyramids follow, each divided by 2min of active recovery at 65-70% HRmax, making it a total of 28min.
  Interventions: Other: Continuous Endurance Training; Other: High-intensity interval training
- High-intensity intervall training (Experimental): HIT: 4x4 min intervals at85-95% HRmax divided by 3x3min of active recovery at 60-70% HRmax, making it a total of 25min.
  Interventions: Other: Continuous Endurance Training; Other: Pyramid Training

INTERVENTIONS:
Other: Continuous Endurance Training — Endurance training with constant work load 31min at 65-75% Hrmax
  Arms: High-intensity intervall training; Pyramid Training
Other: Pyramid Training — One pyramid consists of 8 one-minute blocks. Those are grouped starting with one block of 70-75% HRmax, followed by one block at 75-80% HRmax and another one at 80-85% HRmax. The top of the pyramid are 2 blocks of 85-90% HRmax. Intensity is lowered afterwards with one block of 80-85% HRmax, followed by one block at 75-80% HRmax and last one at 70-75% HRmax. Two more pyramids follow, each divided by 2min of active recovery at 65-70% HRmax, making it a total of 28min.
  Arms: Continuous Endurance training; High-intensity intervall training
Other: High-intensity interval training — HIT: 4x4 min intervals at85-95% HRmax divided by 3x3min of active recovery at 60-70% HRmax, making it a total of 25min.
  Arms: Continuous Endurance training; Pyramid Training

SUMMARY:
It is the aim of our study to compare the effects of 6 and/or 2 years of either HIT (carried out at correctly assessed 85-95% of maximal heart rate), pyramid, or continuous endurance training, on changes of physical exercise capacity in cardiac patients.

DETAILED DESCRIPTION:
The three exercise arms (isocaloric) are composed as follows:

Endurance training: 31 min at 65-75% HRmax, making it a total of 25min; HIT: 4x4min intervals at 85-95% HRmax divided by 3x3min of active recovery at 60-70% HRmax, making it a total of 25 min; Pyramid: One pyramid consists of 8 one-minute blocks. Those are grouped starting with one block of 70-75% HRmax, followed by one block at 75-80% HRmax and another one at 80-85% HRmax. The top of the pyramid are 2 blocks of 85-90% HRmax. Intensity is lowered afterwards with one block of 80-85% HRmax, followed by one block at 75-80% HRmax and last one at 70-75% HRmax. Two more pyramids follow, each divided by 2min of active recovery at 65-70% HRmax, making it a total of 28min.

All protocols are initiated by 5min of warm-up and end with 5min of cool-down, both at 60-70% HRmax.

Primary Outcome: Individual maximum power output in watt (Pmax). Secondary Outcome: Change of power output in watt at lactate tresholds at 2 and 4mmol/l.

ELIGIBILITY:
Inclusion Criteria:

* acute coronary syndrome (STEMI - NONSTEMI)
* aortocoronary bypass surgery
* percutaneous coronary intervention (PCI)
* state after stable coronary heart disease
* state after heart surgeries
* state after myo-, endo-, or pericarditis
* state after heart- or lung-transplantation
* state after heart failure
* state after pulmonary hypertension
* state after peripheral venous disease
* state after electrophysiological surgery
* state after implantation of an implantable cardioverter or difibrillator
* Patients at high risk
* Patients with cardiac dysrhythmias or sudden death

Exclusion Criteria:

* unstable angina pectoris
* Heart failure (NYHA IV)
* acute myo-, endo-, or pericarditis or other infections
* pulmonary-arterial embolism or phlebothrombosis within 6 months
* hemodynamic instable dysrhythmias
* hypertrophic cardiomyopathy
* medical conditions which prevent patients from complying with the exercise program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-01; Primary Completion 2018-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Physical work capacity (PWC) | 6 weeks or 36 weeks
  PWC will be measured by graded exercise testing on cycle ergometer.

SECONDARY OUTCOMES:
Heart rate | 6 weeks or 36 weeks
  Heart rate will be measured by graded exercise testing on cycle ergometer.
Blood pressure | 6 weeks or 36 weeks
  Blood pressure will be measured by graded exercise testing on cycle ergometer.
Lactate Thresholds | 6 weeks or 36 weeks
  Lactate thresholds will be measured by graded exercise testing on cycle ergometer.
Metabolical and cellular blood parameter | 6 weeks or 36 weeks
  Blood will be taken before and after intervention
BMI | 6 weeks or 36 weeks
  BMI will be taken before and after intervention
Gene expression | 6 weeks or 36 weeks
  Gene expression will be taken before and after intervention
Quality of Life | 6 weeks or 36 weeks
  Quality of Life will be taken before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Josef Niebauer, M.D, PhD,MBA, Principal Investigator — Department of Sports Medicine, Prevention and Rehabilitation Paracelsus Medical University
Locations (1):
- Department of Sports Medicine, Prevention and Rehabilitation Paracelsus Medical University, Salzburg, Austria

REFERENCES:
- [Derived] Mayr B, Muller EE, Schafer C, Droese S, Schonfelder M, Niebauer J. Exercise-induced changes in miRNA expression in coronary artery disease. Clin Chem Lab Med. 2021 May 12;59(10):1719-1727. doi: 10.1515/cclm-2021-0164. Print 2021 Sep 27. PMID 33977686
- See also: Paracelsus Medical University Salzburg, Austria — http://www.pmu.ac.at
- See also: Department of Sports Medicine, Prevention and Rehabilitation Paracelsus Medical University — http://www.salk.at/sportmedizin.html
- See also: Salzburg Regional Hospital — http://www.salk.at/